CLINICAL TRIAL: NCT06418750
Title: Evaluation of a Range of Dermo-cosmetic Products to Treat Skin and Nail Toxicity Linked to Bispecific Anti-GPRC5D Bispecific Antibodies in Multiple Myeloma Patients". Myeloma.
Brief Title: Evaluation of a Range of Dermo-cosmetic Products to Treat Skin and Nail Toxicity Linked to Bispecific Anti-GPRC5D Bispecific Antibodies in Multiple Myeloma Patients". Myeloma". Descriptive Pilot Study
Acronym: DELICATESSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC23_0530
Record Dates: First submitted 2024-04-24; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Myeloma Multiple
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Two groups studied: preventive and curative.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group preventive (Other)
  Interventions: Other: dermo-cosmetic product
- group curative (Other)
  Interventions: Other: dermo-cosmetic product

INTERVENTIONS:
Other: dermo-cosmetic product — For patients in the preventive group, treatment with hand serum, gloves/slippers and fortifying solution/dissolving oil will be started on the day of the first administration of Ac bispecific. In the curative group, treatment will begin on inclusion in the study and will be adapted to the lesions present on D0. Treatment will be readjusted on a weekly basis according to the lesions present at the time of the follow-up visit.

SUMMARY:
The aim of this study is to assess the efficacy of range of dermo-cosmetic products (hand/feet serum, nail strengthening solution nail strengthening solution, dissolving oil and gloves/slippers) based on natural products and designed for cancer patients)on bispecific Ac-induced skin and nail toxicity in MM patients treated with anti-CD3xGPRC5D bispecific antibodies.

The effects of supportive care products will be studied as a preventive measure in patients starting treatment with bispecific Ac and as a curative measure in patients undergoing treatment.

Patients will be able to apply the products directly at home according to the study schedule, and a skin and nail toxicity skin and nail toxicity will be performed each time the patient comes for administration of bispecific Ac. Follow-up will be for a total of 6 months (or less if progression occurs earlier), and patients will be asked to complete a quality-of-life questionnaire at protocol inclusion and after 1 month and 6 months of supportive care.

ELIGIBILITY:
Inclusion Criteria:

1. MM patient.
2. Patient starting anti-GPRC5D bispecific Ac therapy OR patient undergoing anti-GPRC5D bispecific Ac therapy with NCI-NCTCAE V5.0 grade ≥2 skin and nail toxicity.
3. Patient with written consent.

Exclusion Criteria:

1. Patients treated or considering treatment with dermatological drugs (dermocorticoids) normally used for hand-foot syndrome OR dermo-cosmetic products (serum or reparative solutions) other than those tested.
2. Patients with atomic dermatitis (eczema)
3. Patients allergic to one or more components of the products tested.
4. Pregnant or breast-feeding women.
5. Patients who are minors or under legal protection (guardianship or safeguard of justice).
6. Patient not affiliated to a social security scheme.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cutaneous and nail toxicity (pain, pruritus, erythema, edema, xerosis, hyperkeratosis, desquamation and onychodystrophy) within one month of starting to use support products. | 1 month
  To evaluate the efficacy of a range of dermo-cosmetic products in preventing/limiting cutaneous and nail toxicity induced by anti-GPRC5D bispecific Ac in MM patients according to the NCI-CTCAE V5.0 scale.

SECONDARY OUTCOMES:
Cutaneous and nail toxicity (pain, pruritus, erythema, edema, xerosis, hyperkeratosis, desquamation and onychodystrophy) occurring after 6 months (or earlier if progression) of use of support products. | 6 month
  To evaluate the efficacy of a range of dermo-cosmetic products in preventing/limiting cutaneous and nail toxicity induced by anti-GPRC5D bispecific Ac in MM patients according to the NCI-CTCAE V5.0 scale.
Total DLQI score after 1 month and 6 months (or earlier if progression) post use of support products. | 1 month/6 month
Pain score after 1 month and 6 months (or earlier if progression) post use of support products. | 1 month/6 month
Satisfaction at 6 months (or earlier if progression) assessed on a Likert scale by the doctor and patient, for each product in the range tested. | 6 month